CLINICAL TRIAL: NCT06415227
Title: Vericiguat in Vasospastic Angina
Brief Title: The Impact of Vericiguat on Microvascular Function in Patients with Documented Vasospastic Angina Pectoris
Acronym: ViVA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jan J. Piek, MD, PhD, Prof. dr., Amsterdam University Medical Center (UMC), Location Academic Medical Center (AMC)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT 2022-502998-42-00
Record Dates: First submitted 2024-04-25; First posted 2024-05-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Vasospastic Angina
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat (2.5 mg, 5 mg and 10 mg) first; placebo second (Experimental): Treatment with Vericiguat will be uptitrated every two weeks to the highest tolerated dose, with a target maintenance dose of maximum 10 mg once daily. After a washout period of 2 weeks, matching placebo will be started and is uptitrated every two weeks to maintain double blinding.
  Interventions: Drug: Vericiguat
- Placebo first; Vericiguat (2.5 mg, 5 mg and 10 mg) second (Placebo Comparator): Matching placebo is uptitrated every two weeks to maintain double blinding. After a washout period of 2 weeks, treatment with Vericiguat will be started and is uptitrated every two weeks to the highest tolerated dose, with a target maintenance dose of maximum 10 mg once daily.
  Interventions: Drug: Vericiguat

INTERVENTIONS:
Drug: Vericiguat — The target dose of vericiguat is 10 milligrams once daily, which will be started at 2.5mg once daily and uptitrated every two weeks to reach the target dose. Dose modification will depend on mean sitting systolic blood pressure and the absence of symptoms indicative of hypotension. The intention of the protocol is to reach and maintain the target study drug dose after completion of uptitration. If the dose is temporarily interrupted, then resumption of study drug treatment and continued uptitration will be considered at any subsequent visit when the investigator feels it is medically appropriate. Vericiguat will be taken orally once daily at about the same time.
  Other Names: Verquvo

SUMMARY:
Vasospastic angina is increasingly recognized as an important contributor to anginal symptoms in patients with non-obstructive coronary artery disease (ANOCA). Endothelial dysfunction and smooth muscle cell dysfunction are considered elementary in the development of vasospastic angina. As one of many functions, the vascular endothelium regulates local vascular tone, mainly through the vasodilatory effect of endothelium-derived nitric oxide (NO). Vericiguat is a soluble guanylate cyclase (sGC) stimulator and thereby acts directly on the NO signalling pathway from the endothelium towards the vascular smooth muscle cells. As such, Vericiguat potentially has an beneficial therapeutic effect in patients with vasospastic angina.The VIVA study aims to demonstrate the effect of Vericiguat on endothelial function and microvascular vasodilator responses, as well as its tolerability and safety in patients with vasospastic angina as the pathophysiological substrate of ANOCA.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Recurrent angina symptoms provoked by exercise and/or repeated attacks of angina at rest at least once weekly despite current medical treatment.
* Absence of (co-existing) flow-limiting coronary artery stenosis (as defined by any coronary artery diameter reduction >50%, or fractional flow reserve≤0.80, or instantaneous wave-free ratio/resting full cycle ratio ≤0.89).
* Unambiguous epicardial and/or microvascular coronary vasospasm according to the COVADIS criteria, documented by invasive acetylcholine provocation testing.
* A female participant is eligible to participate if at least one of the following conditions applies: Women with a confirmed post-menopausal state (defined as amenorrhea for at least 12 months without an alternative medical cause); or premenopausal women with documented hysterectomy, documented bilateral salpingectomy or documented bilateral oophorectomy; or for women of childbearing potential: Negative highly sensitive urine or serum pregnancy test within 24 hours the first dose of study intervention and practicing a highly effective birth control method (failure rate of less than 1%) during the study intervention period / and for at least one month after the last dose of study intervention: progestogen-only subdermal contraceptive implant, intrauterine system (progestin releasing intrauterine device), non-hormonal intrauterine device, bilateral tubal occlusion, azoospermic partner (vasectomized or secondary to medical cause) or heterosexual abstinence.

Exclusion Criteria:

* Impaired left ventricular function (LVEF<50%)
* Significant valvular pathology
* Contraindication for treatment with sublingual nitrates as background medication only, at the discretion of the treating cardiologist.
* Contraindications for treatment with vericiguat: resting systolic blood pressure<100mmHg, severe renal impairment (estimated glomerular filtration rate <15ml/min), severe hepatic impairment.
* Known hypersensitivity to the active substance or to any of the excipients (Microcrystalline cellulose, croscarmellose sodium, hypromellose 2910, lactose monohydrate, magnesium stearate, sodium laurilsulfate).
* Concomitant use of other soluble guanylate cyclase (sGC) stimulators, such as riociguat.
* Concomitant use PDE5 inhibitors, such as sildenafil.
* Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Patients who are pregnant or nursing and those who plan pregnancy in the period up to 1 month after the study;
* Patients with a limited life expectancy less than one year;
* Patients unable to provide written informed consent, or are otherwise not suitable for inclusion according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Microvascular function assessed with LASCA : Area under the curve for cutaneous microvascular conductance during acetylcholine iontophoresis | 10-week and 22-week follow-up
  Difference in area under the curve for cutaneous microvascular conductance in APU/s during acetylcholine iontophoresis after 10-week placebo- versus 10-week vericiguat treatment periods

SECONDARY OUTCOMES:
Microvascular function assessed with LASCA : Peak cutaneous microvascular conductance during acetylcholine iontophoresis | 10-week and 22-week follow-up
  Difference in peak cutaneous microvascular conductance in APU/mmHg during acetylcholine iontophoresis after 10-week placebo- versus 10-week vericiguat treatment periods
Microvascular function assessed with LASCA : Absolute and relative change in cutaneous microvascular conductance (peak-baseline) during acetylcholine iontophoresis. | 10-week and 22-week follow-up
  Difference in the absolute and relative change in cutaneous microvascular conductance from baseline conditions to peak conductance during acetylcholine iontophoresis in APU/mmHg after 10-week placebo- versus 10-week vericiguat treatment.
Vasodilator function assessed with EndoPAT. | 10-week and 22-week follow-up
  Difference in vasodilator function assessed with EndoPAT after 10-week placebo versus 10-week vericiguat treatment expressed by the Reactive hyperemia index (RHI), calculated as the index of signal amplitude pre-to-post occlusion in the occluded arm, divided by the same ratio in the control arm.
Microvascular function assessed with LASCA on placebo versus vericiguat treatment using SNP and insulin. | 10-week and 22-week follow-up
  Difference in cutaneous microvascular conductance in APU/mmHg during SNP or insulin iontophoresis after 10-week placebo- versus 10-week vericiguat treatment periods
Microvascular function assessed with LASCA on placebo versus vericiguat treatment using SNP and insulin. | 10-week and 22-week follow-up
  Difference in the area under the curve for cutaneous microvascular conductance in APU/s during SNP or insulin iontophoresis after 10-week placebo- versus 10-week vericiguat treatment periods
Microvascular function assessed with LASCA stratified by the vericiguat dose reached during the treatment | 10-week and 22-week follow-up
  Difference in peak cutaneous microvascular conductance in APU/mmHg after 10-week placebo versus 10-week vericiguat treatment stratified by the vericiguat dose reached during the treatment phase (5 or 10mg).
Microvascular function assessed with LASCA stratified by the vericiguat dose reached during the treatment | 10-week and 22-week follow-up
  Difference in area under the curve for cutaneous microvascular conductance in APU/s after 10-week placebo versus 10-week vericiguat treatment stratified by the vericiguat dose reached during the treatment phase (5 or 10mg).
Microvascular function assessed with LASCA stratified by the vericiguat dose reached during the treatment | 10-week and 22-week follow-up
  Difference in absolute and relative changes in cutaneous microvascular conductance in APU/mmHg after 10-week placebo versus 10-week vericiguat treatment stratified by the vericiguat dose reached during the treatment phase (5 or 10mg).
Vasodilator function assessed with EndoPAT stratified by the vericiguat dose reached during the treatment | 10-week and 22-week follow-up
  Difference in reactive hyperemia index (RHI) after 10-week placebo versus 10-week vericiguat treatment stratified by the vericiguat dose reached during the treatment phase (5 or 10mg). RHI is calculated as the index of signal amplitude pre-to-post occlusion in the occluded arm, divided by the same ratio in the control arm.
Microvascular function assessed with LASCA stratified by epicardial or microvascular vasospasm endotype. | 10-week and 22-week follow-up
  Difference in peak cutaneous microvascular conductance in APU/mmHg after 10-week placebo versus 10-week vericiguat treatment stratified by epicardial or microvascular vasospasm endotype.
Microvascular function assessed with LASCA stratified by epicardial or microvascular vasospasm endotype. | 10-week and 22-week follow-up
  Difference in area under the curve for cutaneous microvascular conductance in APU/s after 10-week placebo versus 10-week vericiguat treatment stratified by epicardial or microvascular vasospasm endotype.
Microvascular function assessed with LASCA stratified by epicardial or microvascular vasospasm endotype. | 10-week and 22-week follow-up
  Difference in absolute and relative changes in cutaneous microvascular conductance in APU/mmHg after 10-week placebo versus 10-week vericiguat treatment stratified by epicardial or microvascular vasospasm endotype.
Vasodilator function assessed with EndoPAT stratified by epicardial or microvascular vasospasm endotype. | 10-week and 22-week follow-up
  Difference in reactive hyperemia index (RHI) after 10-week placebo versus 10-week vericiguat treatment stratified by epicardial or microvascular vasospasm endotype. RHI is calculated as the index of signal amplitude pre-to-post occlusion in the occluded arm, divided by the same ratio in the control arm.
Quality of life between vericiguat treatment and placebo | 10-week snd 22-week follow-up
  Difference in quality of life measured by the ORBITA-2 application after 10-week placebo versus 10-week vericiguat treatment periods.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by the Seattle Angina Questionnaire (SAQ) Summary Score after 10-week placebo versus 10-week vericiguat treatment periods. The SAQ summary score ranges from 0 to 100 with higher scores indicating less angina, fewer functional limitations, and better quality of life.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by the Rose Dyspnea Score after 10-week placebo versus 10-week vericiguat treatment periods. The Rose Dyspnea Scale is a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by EQ-5D-5L (EuroQol - 5 dimensions - 5 levels. A self-assessed, health-related, quality of life questionnaire) scores after 10-week placebo versus 10-week vericiguat treatment periods. The five severity levels in the EQ-5D-5L are 'no problems', 'slight problems', 'moderate problems', 'severe problems' and 'unable to/extreme problems'.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by the EQ visual analogue scale (EQ-VAS) scores after 10-week placebo versus 10-week vericiguat treatment periods. The EQ VAS component contains a scaled vertical line ranging from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine') where respondents rate their overall health status.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by iPCQ (iMTA (Institute for Medical Technology Assessment) Productivity Cost Questionnaire) index score after 10-week placebo versus 10-week vericiguat treatment periods. The scoring of the iPCQ questionnaire involves three modules assessing productivity losses due to absenteeism (1), presenteeism (2), and productivity losses associated with unpaid work (3). Scores are calculated in costs with a higher score indicating higher productivity loss.
Quality of life between vericiguat treatment and placebo | 10-week and 22-week follow-up
  Difference in quality of life measured by iMCQ (iMTA (Institute for Medical Technology Assessment) Medical Consumption Questionnaire) index score after 10-week placebo versus 10-week vericiguat treatment periods. The scoring of the iMCQ questionnaire involves calculating medical consumption by assessing respondents' answers to relevant questions, which inquire about various forms of care and the frequency of their utilization. A higher score indicates higher health care consumption.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change in quality of life measured by the ORBITA-2 application from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change in quality of life measured by the Seattle Angina Questionnaire (SAQ) Summary Score from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods. The SAQ summary score ranges from 0 to 100 with higher scores indicating less angina, fewer functional limitations, and better quality of life.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change of quality of life measured by the Rose Dyspnea Score from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods. The Rose Dyspnea Scale is a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change of quality of life measured by the EQ-5D-5L (EuroQol - 5 dimensions - 5 levels. A self-assessed, health-related, quality of life questionnaire) scores from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods.The five severity levels in the EQ-5D-5L are 'no problems', 'slight problems', 'moderate problems', 'severe problems' and 'unable to/extreme problems'.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change of quality of life measured by the EQ visual analogue scale (EQ-VAS) scores from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods.The EQ VAS component contains a scaled vertical line ranging from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine') where respondents rate their overall health status.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change of quality of life measured by the iPCQ (iMTA (Institute for Medical Technology Assessment) Productivity Cost Questionnaire) index score from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods. The scoring of the iPCQ questionnaire involves three modules assessing productivity losses due to absenteeism (1), presenteeism (2), and productivity losses associated with unpaid work (3). Scores are calculated in costs with a higher score indicating higher productivity loss.
Quality of life between baseline and end of treatment | 10-week and 22-week follow-up
  Difference in the change of quality of life measured by the iMCQ (iMTA (Institute for Medical Technology Assessment) Medical Consumption Questionnaire) index score from baseline (prior to randomization) to 10-week placebo and 10-week vericiguat treatment periods. The scoring of the iMCQ questionnaire involves calculating medical consumption by assessing respondents' answers to relevant questions, which inquire about various forms of care and the frequency of their utilization. A higher score indicates higher health care consumption.
Angina burden | 10-week and 22-week follow-up
  Angina burden calculated by the frequency of angina attacks for placebo versus vericiguat treatment periods
The occurrence of major adverse cardiac events | 24 weeks
  The occurrence of major adverse cardiac events (hospitalization for angina, spontaneous myocardial infarction, unplanned revascularization, death) during the study period.

OTHER OUTCOMES:
Relationship between vericiguat plasma concentrations and change in microvascular function | 10-week and 22-week follow-up
  Relationship between vericiguat plasma concentrations and change in microvascular function from baseline to 10-week placebo and 10-week vericiguat treatment (in case an overall clinical benefit has been demonstrated).

IPD SHARING:
Plan to Share IPD: Undecided